CLINICAL TRIAL: NCT05744232
Title: The Impact of Low-energy totAl Diet Replacement With Behavioural Support for remIssion of Type 2 DIAbetes on disordEred eatiNg: the ARIADNE Randomised Non-inferiority Controlled Trial
Brief Title: ARIADNE: A Study of Weight Loss for Diabetes Treatment and Wellbeing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R82152/RE004
Record Dates: First submitted 2023-01-25; First posted 2023-02-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-08

CONDITIONS: Type2diabetes; Disordered Eating; Obesity; Overweight and Obesity; Diet Habit
MeSH Terms: conditions — Obesity; Overweight; Feeding Behavior

STUDY DESIGN:
Masking Description: An independent member of the research team, who will not be delivering the intervention or conducting baseline or follow-up assessments, will do the randomisation by inputting the data onto the software. The research team will then notify the participant of their allocation group and further steps.
  Due to the nature of the intervention and the control group, blinding of the participants and the researchers to the intervention is not possible. However, the assessment of the primary outcome will be blinded, as questionnaires will be self-administered online. The PIS will present the study to participants in a more general context, focusing on the impact of total diet replacement on well-being, without mentioning disordered eating, as this could predispose participants in their questionnaire answers and heavily affect the outcomes of this study, introducing measurement bias and weakening the conclusions drawn.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention- Low calorie diet/ Total diet replacement (Experimental): Participants in the intervention group will be offered a dietitian-delivered intervention over 6 months, similar to the NHS pilot of low calorie diets for type 2 diabetes remission. The intervention starts with 12 weeks of low-energy total diet replacement (approx. 860 kcal/day) in a nutritionally replete package of soups, shakes, and bars. It continues with stepped food reintroduction (maximum 6 weeks) as a low-calorie, nutrient-rich diet personalised to the individual participant circumstances and preferences, and weight maintenance (6 weeks).
  Interventions: Behavioral: Low calorie total diet replacement
- Control- usual care (Other): Participants allocated to the control group will be offered and continue benefiting from standard care. Participants will not be stopped from pursuing any behavioural weight management programme but if they do, this will be recorded. Participants will be offered an invitation to a 30-45' 1:1 session with the research dietitian at the end of the study to provide help and signposting as required for the management of their diabetes.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Low calorie total diet replacement — Summary
  1. Weeks 1-12: TDR phase
  2. Weeks 13-14: Food reintroduction phase I
  3. Weeks 15-16: Food reintroduction phase II
  4. Weeks 17 till 20: Food reintroduction phase III
  5. Weeks 21 till 24: Maintenance phase
  Arms: Intervention- Low calorie diet/ Total diet replacement
Other: Usual care — Participants allocated to the control group will be offered and continue benefiting from standard care. Participants will not be stopped from pursuing any behavioural weight management programme but if they do, this will be recorded.
  Arms: Control- usual care

SUMMARY:
The NHS has started a trial-run of a weight loss programme replacing food with 800-calorie shakes and soups for 3 months, offered to people with newly diagnosed type 2 diabetes (T2D) to lose weight and put their diabetes into remission. Some healthcare professionals and charities are sceptical about the programme's effect on people's mental health. They fear it may trigger people to have a negative relationship with food (disordered eating). Some studies show indirectly that these programmes are somewhat safe; however it is not known for sure if it could affect people's relationship with food for the worse. Investigators will invite 56 people with T2D and disordered eating (picked up by questionnaires they will fill in) to participate in a trial. Of these participants, 28 will get TDR and the rest will get their standard care. Investigators will then measure how their scores of disordered eating change at 1, 3, 4, 6, 12 and 24 months. Investigators also plan to analyse the recorded sessions to better understand participants' experiences using TDR and their thoughts about eating and body image. This study will help shed light on how safe this type of diet is for people with disordered eating. It may lead to screening for eating disorders if TDR becomes standard care. If concerns are unfounded, it can reassure people with type 2 diabetes and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent, can communicate in English
* Age between 18 and 65 years inclusive
* Live in England
* BMI ≥27 kg/m2 or higher (adjusted to ≥25 kg/m2 for people of Black, Asian and minority ethnic origin)
* Diagnosed with T2D within 6 years prior to the day of screening
* Global EDE-Q scores ≥2.67
* To have an HbA1c taken in the last 12 months
* Latest HbA1c ≥43 mmol/mol (6.1%) and ≤87 mmol/mol (10%) if on diabetes medication OR latest hbA1c ≥ 48 mmol/mol (6.5%) and ≤87 mmol/mol (10%), if not on diabetes medication.
* If diagnosed with type 2 diabetes more than 1 year since day of screening, the participant must have attended their GP surgery for monitoring/ diabetes review when last offered
* Commit to continue annual reviews with their GP, even if T2D remission is achieved

Exclusion Criteria:

The participant must not enter the study if ANY of the following apply:

* Current or previous clinical diagnosis of an eating disorder
* Combination of EDE-Q ≥4 AND a CIA score ≥16 at screening
* Currently participating in a structured weight loss programme or self-reporting that they have lost >10% of their body weight in the last 3 months
* Insulin use
* Known kidney disease of stage 3/4/5 or eGFR <60 mls/min/1.73 m2 within the last 12 months
* Active substance use disorder
* Active cancer other than skin cancer
* Known proliferative retinopathy that has not been treated
* Porphyria
* Undergone or is awaiting bariatric surgery
* Myocardial infarction or stroke within previous 6 months
* Severe heart failure defined as equivalent to the New York Heart Association (NYHA) grade 3 or 4
* Active liver disease (not including non-alcoholic fatty liver disease)
* Pregnant, breastfeeding, or planning to become pregnant during the course of the study
* Soy or milk or fish allergy, lactose intolerance, or following a vegan diet
* People currently participating in another study or clinical trial of a CTIMP/non-CTIMP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Global score of disordered eating psychopathology | 24 weeks
  Between group difference in scores of disordered eating psychopathology, as measured by the global score of the self-administered Eating Disorders Examination questionnaire (EDE-Q). Scores range from 0 to 6, with higher scores indicating more severe eating disorders psychopathology.

SECONDARY OUTCOMES:
Global score of disordered eating psychopathology | 4, 12, 16, 52 and 104 weeks
  Between group difference in scores of disordered eating psychopathology, as measured by the global score of the self-administered Eating Disorders Examination questionnaire (EDE-Q). Scores range from 0 to 6, with higher scores indicating more severe eating disorders psychopathology.
Subscales of disordered eating psychopathology | 4, 12, 16, 24, 52 and 104 weeks
  Between group difference in sub-scale scores of disordered eating, assessed by the subscale scores of Eating Disorders Examination questionnaire (EDE-Q): Restraint, Eating concern, Shape concern, Weight concern. Subscale scores reflect the severity of the specific characteristics of disordered eating. Higher scores in each subgroup indicate more severe psychopathology.
Psychosocial impairment | 4, 12, 16, 24, 52 and 104 weeks
  Between group difference in psychosocial impairment, assessed by the self-administered clinical impairment assessment (CIA) questionnaire. The CIA measures the severity of psychosocial impairment due to eating disorder features, and scores range from o to 48, with higher scores indicating more severe impairment.
Weight | 4, 12, 16, 24, 52 and 104 weeks
  Changes between group, assessed by self-weighing

OTHER OUTCOMES:
Changes in medication | 12, 24, 52 and 104 weeks
  Changes in diabetes medication between TDR and control
Changes in quality of life | 12, 24, 52 and 104 weeks
  Between group difference in quality of life, measured by the Problem Areas In Diabetes (PAID) Scale. PAID is used to measure distress related to emotions, treatment, food and social support in living with diabetes. Scores range from 0 to 100, with higher scores indicating higher diabetes distress.
Process evaluation of significant changes in disorder eating psychopathology during the intervention | Through study completion, an average of 2 years
  Qualitative analysis of transcribed sessions with the dietitian in people with significant EDE-Q changes (more than 1 SD)
Safety/ New cases needing referral to specialist services | Through study completion, an average of 1 year
  To examine the safety signals of TDR in people with disordered eating, by collecting the incidence of cases of high suspicion of a new eating disorder, measured by referral of participant to see their GP for further referral to specialist services

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Department of Primary Care Health Sciences, Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsompanaki E, Aveyard P, Park RJ, Jebb SA, Koutoukidis DA. An intensive weight loss programme with behavioural support for people with type 2 diabetes at risk of eating disorders in England (ARIADNE): a randomised, controlled, non-inferiority trial. Lancet Psychiatry. 2025 Jul;12(7):483-492. doi: 10.1016/S2215-0366(25)00126-9. PMID 40506207
- [Derived] Tsompanaki E, Aveyard P, Park RJ, Koutoukidis DA. The impact of low-energy total diet replacement with behavioural support for remission of type 2 diabetes on disordered eating (ARIADNE): Protocol for a non-inferiority randomised controlled trial. Contemp Clin Trials. 2024 Jul;142:107542. doi: 10.1016/j.cct.2024.107542. Epub 2024 Apr 27. PMID 38685400